CLINICAL TRIAL: NCT01161992
Title: P.R.O.G.R.E.S.S.: PSC Resource Of Genetic Risk, Environment and Synergy Studies.
Brief Title: Genomics of Primary Sclerosing Cholangitis (PSC)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Konstantinos N. Lazaridis, M.D., Hepatology Consultant, Mayo Clinic
Other Study IDs: 670-02 PSC
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Primary Sclerosing Cholangitis (PSC)
Keywords: Primary Sclerosing Cholangitis; PSC; Cholestatic Liver Disease
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood sample will be drawn at local facility and sent to Mayo Clinic by mail. Stool sample will be collected and sent back to Mayo Clinic by mail. All study related charges will be charged to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: Genetic Analysis — Perform Genome Wide Association Studies.

SUMMARY:
Primary Sclerosing Cholangitis (PSC) is a progressive liver disorder of unknown cause. Current evidence suggests that genes, the genetic material we inherit from our parents, in combination with environmental factors, likely play an important role in the development of PSC.

This study is being done to investigate whether genes make people more likely to develop PSC. Discovery of these genes will help us to better understand how PSC developes and subsequently, to apply new approaches for its prevention, diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men, Women, and Children between the ages of 5-90 with a history of PSC.
* PSC patients who have had a liver transplant are eligible.
* Family members (1st degree relatives) of enrolled PSC patients are eligible.

Exclusion Criteria:

* Individuals with no history of PSC or those unable to provide consent.

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who are patients at Mayo Clinic and are seen in the department of Gastroenterology and Hepatology are recruited by mail and carry a diagnosis of Primary Sclerosing Cholangitis (PSC). Subjects who are not Mayo Clinic patients are encouraged to contact the study coordinator by phone or email to request enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2002-03; Primary Completion 2025-07 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Mapping of Susceptibility Genes in Adult Chronic Cholestatic Liver Diseases
  Adult chronic cholestatic liver diseases, such as Primary Sclerosing Cholangitis (PSC), are progressive liver disorders of unknown cause. Current evidence suggests that genes, the genetic material we inherit from our parents, in combination with environmental factors, likely play an important role in the development of PSC.
  This study is being done to investigate whether genes (the inherited genetic material passed from parents to their children) make people more likely to develop PSC. Discovery of these proposed genes will help us to better understand how PSC progresses,

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos N Lazaridis, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juran BD, Atkinson EJ, Schlicht EM, Larson JJ, Ellinghaus D, Franke A, Lazaridis KN. Genetic polymorphisms of matrix metalloproteinase 3 in primary sclerosing cholangitis. Liver Int. 2011 Jul;31(6):785-91. doi: 10.1111/j.1478-3231.2010.02420.x. Epub 2010 Dec 7. PMID 21134112